CLINICAL TRIAL: NCT03569267
Title: A Phase 1, Single Center, Placebo-controlled, Interventional Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profiles in Healthy Subjects Compared to Placebo
Brief Title: A Study to Evaluate Safety and PK Profiles of OLX10010 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Olix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OLX10010-01
Record Dates: First submitted 2018-05-20; First posted 2018-06-26 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Cicatrix, Hypertrophic
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OLX10010 (Experimental): OLX10010, an siRNA therapeutic, with four different doses by Groups (dose ascending manner with 1, 4, 10, 20 mg)
  Interventions: Drug: OLX10010
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OLX10010 — A cell penetrating asymmetric siRNA (cp asiRNA)
  Arms: OLX10010
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The Study Drug is an investigational drug which is being developed by OliX Pharmaceuticals Inc., with an aim to help people who develop hypertrophic scars (a type of permanent scar) in the future. Hypertrophic scars are formed when a wound becomes red, raised, and itchy before it eventually heals. These scars tend to develop due to disease, surgical operations, or burns. Available physical treatment methods to remove scars include surgery or laser therapy; however these are often accompanied by further complications including pain and recurrence of the scar and can be costly. Similarly, therapeutic agents such as ointments or oral drugs have little to no effect in preventing or treating hypertrophic scars. The aims of this Study are to determine the safety of the Study Drug and any side effects that might be associated with it, and how much of the Study Drug gets into the bloodstream and how long it takes the body to remove it.

The healthy adult subjects can participate in this study in the age between 18 and 60 years old in the UK.

This study will be conducted in 2 parts, Part A and B. Part A will be a single subcutaneous or intradermal dose, dummy controlled study. Part B will be a multiple intradermal dose, dummy controlled study.

DETAILED DESCRIPTION:
The aims of this Study are to determine the safety of the Study Drug and any side effects that might be associated with it, and how much of the Study Drug gets into the bloodstream and how long it takes the body to remove it.

As the selection criteria for the subjects, the healthy adult subjects can participate in this study in the age between 18 and 60 years old in the UK. Both female and male subjects can participate in this study.

This study will be conducted in 2 parts, Part A and B. Part A will be a single subcutaneous dose (Groups A1 to A4) or intradermal dose (Groups A5 to A8), dummy controlled study. Overall, 32 subjects will be studied in 8 groups; 4 groups (Groups A1 to A4) of 4 subjects to assess OLX10010 administered subcutaneously and 4 groups (Groups A5 to A8) of 4 subjects to assess OLX10010 administered intradermally.

Part B will be a multiple intradermal dose, dummy controlled study. Overall, 12 subjects will be studied as 3 groups (Groups B1 to B3) with each group consisting of 4 subjects. In each group, 3 subjects will receive OLX10010 and 1 subject will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, of any race, between 18 and 60 years of age, inclusive, at Screening.
* Body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive, at Screening.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead ECG, vital sign measurements, and clinical laboratory evaluations (congenital non haemolytic hyperbilirubinaemia [eg, Gilbert's syndrome] is not acceptable) at Screening and/or Check in as assessed by the Investigator (or designee).
* Female subjects will be non pregnant and non lactating.
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Exclusion Criteria:

* Male subjects who do not agree, or whose partners of childbearing potential do not agree, to use a male barrier method of contraception (ie, a male condom with spermicide) in addition to a second method of acceptable contraception used by their female partners or to refrain from donating sperm from Check in until 90 days after the Follow up Visit .
* Female subjects of childbearing potential who do not agree to use a highly effective method of birth control in conjunction with male barrier method contraception (ie, a male condom with spermicide) or to refrain from donating ova from the time of signing the ICF until 90 days after the Follow up Visit.
* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
* Subjects with serum creatinine >ULN.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
* History of alcoholism or drug/chemical abuse within 2 years prior to Check in.
* Alcohol consumption of >28 units per week for males and >21 units for females. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1⁄6 gill (25 mL) of spirits.
* Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) at Screening and/or Check in.
* Positive hepatitis panel and/or positive human immunodeficiency test at Screening. Subjects whose results are compatible with prior immunisation and not infection may be included at the discretion of the Investigator.
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 3 months (or 5 half lives, whichever is longer) prior to Check in.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-related adverse events as assessed by CTCAE v4.0 | Day 14 (single dose)
  Incidence and severity of adverse events; vital sign measurements; 12-lead electrocardiogram (ECG) parameters; incidence of clinical laboratory abnormalities, based on haematology, clinical chemistry, and urinalysis test results; analysis of coagulation parameters; physical examinations; local tolerability assessments of subcutaneous and intradermal injection sites

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, Dr., Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit (CRU) Ltd., Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Ethics Review Panel. Requestors will be required to sign a Data Access Agreement.